CLINICAL TRIAL: NCT03450512
Title: Incidence of Neutropenic Enterocolitis Study in Acute Myeloid Leukemia Patients During Intensive Therapy (DECLAM).
Brief Title: Incidence of Neutropenic Enterocolitis Study in Acute Myeloid Leukemia Patients During Intensive Therapy
Acronym: DECLAM
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0031
Record Dates: First submitted 2018-02-05; First posted 2018-03-01 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Neutropenic enterocolitis; Acute myeloid leukemia; Abdominal tomodensitometry
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Enterocolitis, Neutropenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prospective study on digestive affections in an homogeneous cohort of hematological patients — Systematic realization during the induction and/or every consolidation of a CTscan with injection, at the same time as the thoracic CTscan (to research an invasive fungal bronchopulmonary infection), in front of a febrile neutropenia with persistent fever after 5 days of antibiotics and presence of digestive signs.
  Statement of the information characterizing the digestive affection: clinical symptoms, microbiological, characteristic, realized additional explorations, infectious complications and specific therapeutics.
  The abdominal scanner will be repeated in case of suspicion of complication or clinical worsening. In case of EC, the abdominal scanner will be realized before beginning the next cycle of AML treatment to evaluate digestive remission. Finally, a CT scan, will be performed when digestive disease, digestive neoplasia or digestive symptoms are noted at AML diagnosis.

SUMMARY:
Neutropenia after induction or consolidation therapy for acute myeloid leukemia (AML) patients is associated with a high morbi-mortality rates, especially due to infectious complications. These are managed according to international recommandations (ECIL and IDSA) with antibiotherapy and antifungal strategy. Although the patients suffer of digestive symptoms, intestinale complications are really less explored. Neutropenic enterocolitis (NE), cytomegalovirus (CMV) colitis, Clostridium difficile colitis, specific lesion, ischemic colitis are not well-known. No prospective study evaluate NE and these digestive complications which have high morbi-mortality rates.

DETAILED DESCRIPTION:
This is the first prospective study on digestive affections in an homogeneous cohort of hematological patients. These affections are unknown in neutropenic patients with digestive symptoms after induction or consolidation courses pour AML although causing high morbi-mortality rates (infections, denutrition, loss of autonomy…).

The aim of the study is to evaluate incidence of NE by clinical signs and with a systematic CT scan performed at day 5 of fever during aplastic period. An early diagnostic could decrease complications and evaluate gravity criteria which could imply surgery therapy.

The physician will performe a CTscan with injection during the induction and/or every consolidation, at the same time as the thoracic CTscan (to research an invasive fungal bronchopulmonary infection), in front of a febrile neutropenia with persistent fever after 5 days of antibiotics and presence of digestive signs.

The clinical, microbiological, radiological symptoms will be registered at every time of febrile neutropenia with digestive symptoms at induction and each consolidation courses. The patient will be get out of the study when the AML is refractory, hematopoietic stem cell transplantation is required or if whenever he want. The last visit will be at the end of consolidation courses.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* inclusion criteria:

Every patient of hematology:

* Able to receive an intensive treatment for AML (induction then intensive consolidations) causing a neutropenia with high infectious risk
* In state to give its consent
* Affiliated to a social security system

Exclusion Criteria:

* The minor patients
* The patients affected by AML not being able to receive an intensive therapy
* The patients affected by acute promyelocytic leukaemia
* The pregnant women
* The patients with HIV, hepatitis B or C
* The patients under guardianship or guardianship or deprived of freedom by a court or administrative order (according to articles L1121-6 and L1121-8 of the Public health code)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with febrile neutropenia after induction or consolidation courses for AML( acute myeloid leukemia ).
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2024-11-11 (Estimated); Study Completion 2024-11-13 (Estimated)

PRIMARY OUTCOMES:
the arisen of EC in the CT scan | 1 day
  The main assessment criteria is the arisen of EC in the CT scan with injection realized at day 5 of fever under antibiotics for every inclusive patient, with febrile neutropenia, and presenting digestive symptoms during the period of aplasie post-chemotherapy after exclusion from the other diagnosis (infectious colitis and other abdominal syndromes).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Amiens-Picardie, Amiens
  - CHU de Caen, Caen
  - Henri Becquerel Center, Rouen